CLINICAL TRIAL: NCT05817539
Title: Early Deresuscitation Strategy Driven by Tissue Perfusion in Renal Replacement Therapy in Patients With Acute Renal Failure in Intensive Care Unit. A Randomized Study
Brief Title: Early Deresuscitation Strategy Driven by Tissue Perfusion in Renal Replacement Therapy in Patients With Acute Renal Failure
Acronym: EarlyDry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 69HCL22_1095
Record Dates: First submitted 2023-04-05; First posted 2023-04-18 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Acute Kidney Injury; Fluid Overload
Keywords: Renal Replacement Therapy (RRT); Ultrafiltration; Deresuscitation; Fluid balance; Fluid overload; Tissue perfusion
MeSH Terms: conditions — Acute Kidney Injury; Edema

STUDY DESIGN:
Who Masked: Participant
Masking Description: For this protocol, the double blind is impossible to set up. Clinicians in charge of patients and implementing the depletion strategy cannot be blinded.
  The patients will be blinded, they will not be aware of strategy applied. The medical staff will ensure that no information about the intervention is given to the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corrective strategy (Experimental): In the experimental group, all patients will have a UFnet settled (2 ml/kg/h ) in order to reach the patient baseline body weight.
  Interventions: Procedure: Fluid balance negativation
- Stabilizing strategy (Other): In the control group, all patients will have a UFnet 2 ml settled (0 to 1 ml/kg/h) in order to stabilize the patient body weight.
  Interventions: Procedure: Body weight Stabilization

INTERVENTIONS:
Procedure: Fluid balance negativation — During the RRT, UFnet will be settled on 2ml/kg/h and adapted to hemodynamic tolerance and tissue perfusion .
  When the patient's baseline body weight is reached the UF net will be settled to maintain it.
  In case of failure of the fluid balance negativation after 24h, UFnet will be settled on 3ml/kg/h. Then when the baseline body weight is reached UFnet will be settled on 0.5 et 1ml/kg/h or if necessary adapted to 1,5ml/kg/h to maintain it
  In case of hemodynamic intolerance (NADN > 0,5 µg/kg/min) or tissue hypoperfusion, UF net will be stopped during 6 hours and restarted if NADN < 0,5 µg/kg/min and without tissue hypoperfusion.
  Arms: Corrective strategy
Procedure: Body weight Stabilization — During the RRT, UFnet will be settled between 0 et 1 ml/kg/h and adapted in case of weight stabilization failure or hemodynamic intolerance.
  In case of weight stabilisation failure ( variation >3% after 24h), the UF net can be increased to 1,5 ml/kg/h, as long as high intakes require UFnette at 1.5mL/kg/h to stabilize water balance, with daily reassessment.
  In case of hemodynamic intolerance (NADN > 0,5 µg/kg/min), UF net will be stopped during 6 hours and restarted if NADN < 0,5 µg/kg/min.
  Arms: Stabilizing strategy

SUMMARY:
In Intensive Care Unit (ICU) patients with acute kidney injury (AKI) and treated with renal replacement therapy (RRT) often present a fluid overload which is associated with morbidity (mechanical ventilation duration increase, kidney recovery decrease) and mortality.

Patients' prognostic could be improved by correcting the fluid overload with net ultrafiltration (UFnet) however it may lead to harmful iatrogenic hypovolemia responsible of deleterious ischemic lesions.

In usual practice, UF net prescription are variable and there are different international recommendations. Some observational studies suggest that using a UFnet between 1 et 1.75 mL/kg/h in fluid overloaded patient decrease mortality.

Fluid overload increases morbidity and mortality, particularly in RRT. Studies without RRT argue for an efficacy of management by decreasing the fluid overload .Cohort studies suggest to use a moderate UFnet instead of a low UFnet. Some data from studies on early versus late RRT that relate the fluid balance or correct the fluid overload during the early strategy argue for a beneficial effect of an early deresuscitation strategy

Consequently, the impact of a moderate UFnet (to decrease the fluid overload) compared to a low UFnet (to stabilize the fluid overload) in a randomized interventional study could be assessed.

The study hypothesis is that :

an early fluid overload deresuscitation protocol with a high UFnet (2 ml/kg/h) targeting both the negativation of cumulated fluid balance to reach a dry weight and the maintenance of tissue perfusion.

Compared to

fluid overload deresuscitation protocol with a low UFnet (between 0 and 1 ml/kg/h) to reach a stabilization of cumulated fluid balance without monitoring the tissue perfusion.

could improve overall, renal, hemodynamic and respiratory prognosis in fluid overloaded patients with renal replacement therapy in ICU

ELIGIBILITY:
Inclusion Criteria:

1. Acute kidney injury treated by continuous renal replacement therapy in ICU less than 7 days,
2. At least 1 organ failure during ICU in addition to AKI (mechanical ventilation or oxygen therapy or vascular filling > 1000ml or vasopressor exposure > 12 hours),
3. Weight loss of less than 3% since starting a net UF or Cumulative UF net less than 2000ml before inclusion,
4. Norepinephrine < 0,5 µg/kg/min,
5. Absence of hypoperfusion signs defined by the presence of at least 2 out of 4 criteria:

   * TRC > 3s at the finger
   * Marbrure score > 2
   * Lactate > 2 mmol/L
   * ScVO2< 60%,
6. Fluid overload defined as follows :

   * fluid overload > 5% of base weight (based on cumulative fluid balance or a weight gain) and/or
   * Obvious oedema of the lumbar region or flanks (oedema > 1cm bucket depth).

Exclusion Criteria:

1. Chronic renal failure hemodialyzed before admission to the ICU,
2. Mechanical circulatory support (ECMO, LVAD),
3. Pregnant, child -bearing age or lactating women,
4. Stroke based on the combination of central neurological symptoms (aphasia, hemiplegia, hemiparesis) associated with compatible brain imaging, less than 30 days,
5. Intestinal ischemia less than 7 days documented non-operated,
6. Interventional study participation or exclusion period on going,that may interfere with the present study
7. Guardianship, curatorship or safeguard of justice,
8. Absence of signature of free and informed consent by the patient and/or relative,
9. Patients not affiliated to a social security scheme or beneficiaries of a similar scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of organ replacement free-days | Day 30
  Number of organ replacement free-days, i.e, number of renal replacement therapy-free days, number of vasopressor-free days, number of ventilator-free day.
  Number of days between 2 same type organ replacement interruption is not counted.
  In case of death before 30 days, number of days is censored to 0.

SECONDARY OUTCOMES:
Mortality decrease | 30 days
  Number of deaths
Number of renal replacement therapy-free days increase | Day 30
  Number of renal replacement therapy-free days
Number of ventilator-free day increase | Day 30
  Number of ventilator-free day
Number of vasopressor-free day increase | Day 30
  Number of vasopressor-free day
Duration of intensive care unit stay | Up to Day 30
  Number of days in ICU
SOFA score evolution | From Day 0 up to Day 5
  SOFA score : Sepsis-related Organ Failure Assessment, min : 0 max : 24 (worse)
Incidence of arrhythmias and cardiac conduction disorders in both group | From Day 0 up to Day 5
  Number of arrhythmias and cardiac conduction disorders occurrence on ECG
Incidence of intestinal ischemia in both group | From Day 0 to Day 30
  Number of intestinal ischemia on CT scan or endoscopy
Incidence of strokes | From Day 0 to Day 30
  Number of ischemic strokes occurrence on imagery
Incidence of delirium | Between Day 0 and Day 5
  Presence of delirium assessed with the CAM ICU scale : positive or negative score. A positive score means presence of delirium
Renal recovery assessment | Day 30
  Renal recovery is defined according to MAKE 30 scale :
  * Survival
  * Absence of renal replacement therapy
  * Day 30 creatinine level < baseline creatinine x 200 %

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - Centre Hospitalier d'Ajaccio, Ajaccio
  - CHU Amiens-Picardie, Amiens
  - Service d'Anesthesie-Réanimation, Hôpital Louis Pradel, Hospices Civils de Lyon, Bron
  - CHU Caen Normandie, Caen
  - Service de Réanimation, CHU de Dijon, Dijon
  - GHP Saint Joseph Marie Lannelongue, Le Plessis-Robinson
  - CHU Lille - Hôpital Roger Salengro, Lille
  - Hôpital Edouard Herriot, Groupement Hospitalier Centre, Lyon
  - Hôpital de la Croix Rousse, Lyon
  - Service de Réanimation, Clinique de la Sauvegarde, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Département d'anesthésie réanimation Hôpital Européen Georges Pompidou, Paris
  - Hôpitaux de Bradois - CHRU Nancy, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No